CLINICAL TRIAL: NCT03068923
Title: Predicting and Preventing Poor Outcomes of Venous Thromboembolism in Children
Brief Title: Thrombosis Outcomes in Pediatric Venous Thromboembolism
Acronym: TOP
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Ayesha Zia, Associate Professor of Pediatrics, University of Texas Southwestern Medical Center
Other Study IDs: STU 122015-029; 1K23HL132054-01 (NIH)
Record Dates: First submitted 2017-02-22; First posted 2017-03-03 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Venous Thromboembolism
Keywords: Blood clot; Deep Vein Thrombosis; Pulmonary Embolism; Lower Extremity; Upper Extremity; Cerebral sinus; Renal vein; Portal vein; thrombin; fibrinolysis; coagulation; anticoagulation; Post trombotic syndrome; Post pulmonary embolism syndrome; Chronic thromboembolic pulmonary hypertension
MeSH Terms: conditions — Venous Thromboembolism; Thrombosis; Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and DNA samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
'The TOP Study' is a prospective cohort study whose main objective is to develop better prognostic biomarkers and identify children at risk of adverse thrombotic outcomes very early in the course after an initial venous thromboembolic events (VTE). The study will compare biomarkers in children that develop poor VTE outcomes (such as recurrence, postthrombotic syndrome and post PE impairment ) after an initial VTE with those that do not develop such outcomes.

DETAILED DESCRIPTION:
All newly diagnosed patients with a first radiologically confirmed thrombotic event (any site) diagnosed at Children's Medical Center, Dallas will be followed prospectively with global coagulation assessment over a 24-month period, and monitored for development of carefully defined adverse VTE outcomes in a blinded manner. Biomarker assessment will include global coagulation assays (thrombin generation assay and modified thromboelastography to study fibrinolysis) at 3, 6, 12, 18 and 24 months post VTE diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls age birth (0 years) to equal to or less than 21 years
* A radiologically confirmed first venous thromboembolism episode (both extremity and non-extremity) who have completed anticoagulation therapy as per the 9th edition of the ACCP guidelines

Exclusion Criteria:

* Known malignancy
* Pregnancy or immediate post-partum period (12 weeks after delivery)
* Sickle cell disease
* Known bleeding disorder

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Newly diagnosed patients with first venous thromboembolism who have completed therapeutic anticoagulant therapy
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-03-09 (Actual)

PRIMARY OUTCOMES:
Postthrombotic syndrome (PTS) | within 24 months after diagnosis of VTE
  PTS as assessed by the validated Manco-Johnson and the modified Villata PTS instruments determined a priori and confirmed by an endpoint adjudicating committee
Symptomatic recurrent venous thromboembolism | within 24 months after diagnosis of VTE
  Recurrent VTE as assessed by ISTH proposed recurrent VTE clinical criteria
Post-pulmonary embolism (PE) impairment | within 24 months after diagnosis of VTE
  Post-PE impairment, defined as deterioration (compared to discharge or previous follow-up visit), or persistence, in a) echocardiographic parameters of right ventricular (RV) dysfunction (defined by abnormal RV basal diameter or abnormal right atrial end systolic area or abnormal tricuspid annular plane systolic excursion or presence of pericardial effusion) and/or pulmonary hypertension (defined by abnormal estimated right atrial pressure or elevated systolic tricuspid regurgitant velocity), and clinical, functional parameters of RV failure (new appearance of symptoms of heart failure or abnormal six-minute walking distance or elevated brain natriuretic peptide (BNP) plasma levels or abnormal peak O2 uptake on cardiopulmonary exercise testing)

SECONDARY OUTCOMES:
Post-thrombotic sequelae | Within 24 months after diagnosis of VTE
  Site specific sequelae after cerebral sinus venous, portal vein and renal vein thrombosis as assessed by ISTH recommended guidelines
Change in quality of life | Within 24 months after diagnosis of VTE
  Quality of life by PedsQL (TM)

OTHER OUTCOMES:
Change in Physical Activity scores | Within 24 months after diagnosis of VTE
  Physical activity as determined by Gordin questionnaire
Elastic Compression Stocking (ECS) use over time | Within 24 months after diagnosis of VTE
  ECS use will be assessed by ECS log/diary documenting dedicated (use for at least 6 days/week), moderate (use for 4-5 days/week) or poor use (<4 days/week)
Loss of venous access | 12 months post DVT diagnosis
  Loss of venous access in subjects with catheter related DVT of the upper extremity DVT as defined by >30% of the narrowing of the involved vein as assessed by doppler ultrasound or contrast venography
Venous valvular reflux | 12 months post DVT diagnosis
  Venous valvular reflux in subjects with lower extremity DVT will be assessed as present (>0.5 seconds) or absent (<0.5 seconds) at the 12 month post diagnosis visit with a standardized venous reflux ultrasound procedure

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Zia, M.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Children's Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zia A, Russell J, Sarode R, Veeram SR, Josephs S, Malone K, Zhang S, Journeycake J. Markers of coagulation activation, inflammation and fibrinolysis as predictors of poor outcomes after pediatric venous thromboembolism: A systematic review and meta-analysis. Thromb Res. 2017 Dec;160:1-8. doi: 10.1016/j.thromres.2017.10.003. Epub 2017 Oct 7. PMID 29078111